CLINICAL TRIAL: NCT06416384
Title: The Effect of Hand Massage on Post-Dialysis Fatigue and Recovery Time in Hemodialysis Patients
Brief Title: Post-Dialysis Fatigue and Recovery Time in Hemodialysis Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AU-SBE-SA-02
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Hemodialysis; Fatigue; Massage
Keywords: hemodialysis patient; fatique; hand massage; nursing; recovery time
MeSH Terms: conditions — Fatigue | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled, single-blind, experimental study.
Who Masked: Outcomes Assessor
Masking Description: Single-blind (outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand Massage Group (Experimental): The researcher applied a hand massage to the hand area of the patients in the experimental group on the side without fistula for five minutes, three times a week for four weeks.
  Interventions: Other: Control Group
- Control Group (Other): Patients in the control group received routine nursing care in the clinic for four weeks.
  Interventions: Other: Hand Massage Group

INTERVENTIONS:
Other: Hand Massage Group — The patients in the hand massage application group were asked by the researcher; Hand massage with olive oil was applied 12 times in total, three times a week for four weeks. No application was made to the side with fistula.
  Other Names: Experimental
  Arms: Control Group
Other: Control Group — Patients in the control group received routine nursing care in the clinic for four weeks.
  Other Names: Control
  Arms: Hand Massage Group

SUMMARY:
This study aims to examine the effect of hand massage on patients receiving HD treatment on the severity of post-dialysis fatigue and post-dialysis recovery time.

DETAILED DESCRIPTION:
After obtaining the necessary permissions for the research, informing the patients about the purpose, importance and method of the study by the researcher, and having the volunteer patients read and sign a consent form, the patients were randomly divided into two groups. Randomization of the groups was done in a computer environment.

ELIGIBILITY:
Inclusion Criteria:

* Those who are 18 years or older,
* Receiving hemodialysis treatment for at least 3 months,
* Receiving hemodialysis treatment three times a week,
* Does not have any open wounds in the area to be applied,
* No active fistula in the arm to be treated,
* Does not have a hearing impairment,
* Sufficient to understand the questions,
* Open to communication and cooperation,
* Volunteer and willing for research

Exclusion Criteria:

* Having an active oncological problem or receiving oncological treatment,
* Those with health problems that require contact isolation,
* The number of dialysis sessions changed during the study,
* Those who lost their lives while working,
* Those who had a kidney transplant during the study,
* Those who want to leave voluntarily at any stage of the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-11-07 (Estimated)

PRIMARY OUTCOMES:
fatigue severity | one week= first session
  Fatigue severity was evaluated before starting the application (pre-test)
  Post-Dialysis Fatigue Scale: Kodama et al. The "Post-Dialysis Fatigue Scale" developed by (2020) is a five-item likert type scale consisting of 13 items. The scale is used to evaluate the severity of fatigue by examining the factors associated with fatigue observed after the end of treatment in dialysis patients. According to Özen et al. (2021) the total number of items in the scale after Turkish validity and reliability made by is 11.
recovery time | One week= first session
  Recovery time after dialysis was evaluated before starting the application (pre-test)

SECONDARY OUTCOMES:
fatique severity | After 4 weeks
  The effect of hand massage on fatigue severity was measured
  Post-Dialysis Fatigue Scale: Kodama et al. The "Post-Dialysis Fatigue Scale" developed by (2020) is a five-item likert type scale consisting of 13 items. The scale is used to evaluate the severity of fatigue by examining the factors associated with fatigue observed after the end of treatment in dialysis patients. According to Özen et al. (2021) the total number of items in the scale after Turkish validity and reliability made by is 11.
recovery time after dialysis | After 4 weeks
  The effect of hand massage on recovery time after dialysis was measured

CONTACTS AND LOCATIONS:
Overall Officials: Eylem Topbaş, Phd, Study Director — Amasya University; Seyit Ahmet KORKMAZ, Principal Investigator — Amasya University health sciences institute
Locations (1):
- Amasya University İnstitute of Health Sciences, Amasya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It can only be shared after publication upon special request from the authors.